CLINICAL TRIAL: NCT01807871
Title: Treatment of Smoking Lapses and Relapses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Hughes, Faculty Department of Psychiatry, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M12-113; R01CA165080 (NIH)
Record Dates: First submitted 2013-03-04; First posted 2013-03-08 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Smoking Cessation
Keywords: nicotine dependence; smoking cessation; lapse; relapse; tobacco; nicotine patch; nicotine replacement therapy; NRT
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Recurrence | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nicotine patch, experimental use (Experimental): Participants will continue to use nicotine patch after they lapse and resume smoking as long as smoking is less than 75% of pre study levels.
  Interventions: Drug: nicotine patch, experimental use
- nicotine patch, labeled use (Active Comparator): Participants will discontinue using the nicotine patch when they resume smoking. This is the current FDA approved use of the nicotine patches.
  Interventions: Drug: nicotine patch, labeled use

INTERVENTIONS:
Drug: nicotine patch, experimental use — nicotine patch-transdermal, continue during lapses Nicotine patches are used according to normal package label, except if the participant lapses and smokes, they will continue to use the patch.
  Other Names: Nicoderm Clear 21 mg; Nicoderm Clear 14 mg; Nicoderm Clear 7 mg
  Arms: nicotine patch, experimental use
Drug: nicotine patch, labeled use — nicotine patch-transdermal, discontinue during lapses Participants will use the nicotine patch while abstinent, but will remove the patch if there is a lapse and smoking resumes. This is the use indicated on current FDA approved labeling.
  Other Names: Nicoderm Clear 21 mg; Nicoderm Clear 14 mg; Nicoderm Clear 7 mg
  Arms: nicotine patch, labeled use

SUMMARY:
Many smokers who try to stop smoking with nicotine medications (NM) such as gum, lozenge and patch, go back to smoking (i.e., a slip or lapse). Currently, labeling on many NM products tells smokers who lapse while using NM to stop NM. However, some studies suggest it is safe to continue NM upon a lapse and that doing so dramatically increases success at quitting. The investigators will test this by doing a randomized trial in which all treatment and measures are done from home with paper, phone or computer surveys. The investigators will recruit smokers who want to quit, provide them with 10 weeks of nicotine patch treatment and 5 weeks of counseling. One group will be asked to stop use of the patch if they lapse and the other group will be asked to continue use of the patch if they lapse. The investigators will compare the groups on their success at quitting and side-effects.

DETAILED DESCRIPTION:
Objectives:

To test our hypothesis that among the subset of the 770 enrolled participants who quit smoking and then lapsed while using the nicotine patch, those randomized to continue the patch post-lapse will be more likely to be 7-day point prevalent abstinent at 4-month follow-up than those randomized to discontinue the patch post-lapse.

To test whether the amount of patch use post-lapse, craving, withdrawal, cigs/day, motivation to quit, confidence in quitting, nicotine reinforcement from cigarettes, and self-efficacy mediate any effect of post-lapse patch use on abstinence.

To test whether the incidence of adverse events (AEs) during post-lapse patch use is minimal.

Purpose:

Over the counter (OTC) NRT is, by far, the most common treatment for smoking cessation in the United States (Cokkinides, Ward, Jemel, & Thun, 2005). Over 80% of those using OTC NRT will lapse (Stead, Perera, Bullen, Mant, & Lancaster, 2008). One possible reason for this high rate of relapse is that NRT package labeling states "do not use if you continue to smoke", and the majority of smokers believe this means it is best to stop using NRT upon a lapse; e.g., the only survey on real-world use of NRT during a lapse episode found that 77% of smokers discontinued NRT after a lapse (Pierce & Gilpin, 2002). The investigators and others (Bader, McDonald, & Selby, 2009) believe continuing NRT during a lapse episode will a) relieve craving and withdrawal (West & Shiffman, 2001), b) block the reinforcing effects of smoking (Perkins, Fonte, Meeker, White, & Wilson, 2001; Rose & Behm, 2004), c) help smokers smoke less (Hughes & Carpenter, 2005), and d) increase self-efficacy, all of which should help smokers re-establish abstinence.

Study design:

The investigators are proposing a parallel groups randomized controlled trial (RCT) in which all treatment and monitoring occur via phone, and medication via mail. The investigators will recruit about 770 smokers to receive phone counseling before and after the quit date and nicotine patches for 10 weeks after the quit date. At study entry, smokers will be randomized to a "Continue NRT" or a "Discontinue NRT" condition. The Continue NRT participants will be advised that, if they lapse, they should continue NRT. Smokers randomized to the Discontinue NRT condition will be advised that, if they lapse, they should discontinue NRT use. The messages will also include rationales. Messages will be delivered several times via written material, Interactive Voice Response (IVR) messages and during phone counseling. Participants will record cigs/day nightly via a phone-based IVR system for 10 weeks. If the IVR detects a lapse during the first 10 weeks of the study, it will encourage the participant to re-establish abstinence as soon as possible and repeat the condition-appropriate message about post-lapse NRT use. After the 10-week treatment period, the investigators will use monthly questionnaires (online or paper) to assess recent smoking, cigs/day, NRT use, and other stop-smoking medications.

Subject selection:

Men and women, minorities and children over 18 will be included. Pregnant and breastfeeding women, women who plan to become pregnant and those at risk for AEs from NRT will be excluded. Our goal is to recruit a sample of the same gender, ethnicity/race prevalence as that of US smokers interested in quitting; i.e. 52% men, 78% White/Non-Hispanic, 11% Black, 8% Hispanic and 3% other ethnicities/races (Hughes & Callas, 2010). The investigators do not have data on which to estimate the percent who will be children between ages 18-21 but most studies suggest very few young smokers are interested in formal treatment (Sussman, 2002).

Number of subjects:

The investigators have chosen an initial inclusion of 770 smokers to obtain a sample size of 490 smokers who lapse on NRT.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* daily smoker of 10 or more cigarettes per day for at least 1 year
* state they plan to probably or definitely quit smoking in the next month
* have a home or cell phone
* willing to use nicotine patch
* good command of written and spoken English
* weigh at least 100 pounds
* US citizen or permanent resident alien

Exclusion Criteria:

* use of non-cigarette tobacco in the last month
* use of a smoking cessation medication or smoking cessation counseling in the last month
* medical contraindication to use of patch
* other person in household already in our study
* previously a participant in the study
* currently pregnant or breast feeding
* plan to become pregnant in the next 6 months
* regularly works the overnight shift
* use of electronic cigarettes in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Hughes, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cokkinides VE, Ward E, Jemal A, Thun MJ. Under-use of smoking-cessation treatments: results from the National Health Interview Survey, 2000. Am J Prev Med. 2005 Jan;28(1):119-22. doi: 10.1016/j.amepre.2004.09.007. PMID 15626567
- [Background] Stead LF, Perera R, Bullen C, Mant D, Lancaster T. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD000146. doi: 10.1002/14651858.CD000146.pub3. PMID 18253970
- [Background] Pierce JP, Gilpin EA. Impact of over-the-counter sales on effectiveness of pharmaceutical aids for smoking cessation. JAMA. 2002 Sep 11;288(10):1260-4. doi: 10.1001/jama.288.10.1260. PMID 12215133
- [Background] Bader P, McDonald P, Selby P. An algorithm for tailoring pharmacotherapy for smoking cessation: results from a Delphi panel of international experts. Tob Control. 2009 Feb;18(1):34-42. doi: 10.1136/tc.2008.025635. Epub 2008 Oct 9. PMID 18845621
- [Background] West R, Shiffman S. Effect of oral nicotine dosing forms on cigarette withdrawal symptoms and craving: a systematic review. Psychopharmacology (Berl). 2001 May;155(2):115-22. doi: 10.1007/s002130100712. PMID 11400998
- [Background] Perkins KA, Fonte C, Meeker J, White W, Wilson A. The discriminative stimulus and reinforcing effects of nicotine in humans following nicotine pretreatment. Behav Pharmacol. 2001 Feb;12(1):35-44. doi: 10.1097/00008877-200102000-00004. PMID 11270510
- [Background] Hughes JR, Carpenter MJ. The feasibility of smoking reduction: an update. Addiction. 2005 Aug;100(8):1074-89. doi: 10.1111/j.1360-0443.2005.01174.x. PMID 16042638
- [Background] Sussman S. Effects of sixty six adolescent tobacco use cessation trials and seventeen prospective studies of self-initiated quitting. Tob Induc Dis. 2002 Jan 15;1(1):35-81. doi: 10.1186/1617-9625-1-1-35. PMID 19570247
- [Result] Hughes JR, Solomon LJ, Peasley-Miklus CE, Callas PW, Fingar JR. Effectiveness of continuing nicotine replacement after a lapse: A randomized trial. Addict Behav. 2018 Jan;76:68-81. doi: 10.1016/j.addbeh.2017.07.023. Epub 2017 Jul 14. PMID 28756042
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between April 2013 and July 2015
Period: Overall Study
Arm/Group | Nicotine Patch, Experimental Use | Nicotine Patch, Labeled Use
Started | 356 | 345
Completed | 178 | 127
Not Completed | 178 | 218

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Patch, Experimental Use | Nicotine Patch, Labeled Use | Total
Number analyzed (Participants) | 356 | 345 | 701
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11) | 45 (12) | 45 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 207 | 397
  Male | 166 | 138 | 304
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 170 | 179 | 349
  Black Non-Hispanic | 128 | 123 | 251
  Hispanic | 45 | 32 | 77
  Other | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 356 | 345 | 701

OUTCOME MEASURES:

1. Primary Outcome: Point-prevalent Abstinence at 4 Months
Description: To test our hypothesis that among the subset of the 701 enrolled participants who quit smoking and then lapsed while using the nicotine patch, those randomized to continue the patch post-lapse will be more likely to be 7-day point-prevalent abstinent at 4 month follow-up than those randomized to discontinue the patch post-lapse. 7-day point prevalent abstinence was assessed by response to the question "In the last 7 days, on how many days did you smoke" on the 4 month follow-up survey. Respondents who replied "0" were classified as "Yes" for 7-day point-prevalent abstinence; all other responses (including missing) were classified as "No".
Time Frame: 4 months after the quit date
Population: Participants who lapsed while using the nicotine patch
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Patch, Experimental Use | Nicotine Patch, Labeled Use
Number analyzed (Participants) | 178 | 127
Participants | 90 | 59
Statistical Analysis 1: Comparison: Nicotine Patch, Experimental Use vs Nicotine Patch, Labeled Use; Test type: Superiority; p = 0.48, Chi-squared

2. Secondary Outcome: Mediators of Effect of Post-lapse Nicotine Replacement Therapy Use on Abstinence
Description: To test whether the amount of use of nicotine patch post-lapse, craving, withdrawal, cigs/day, motivation to quit, confidence in quitting, nicotine reinforcement from cigarettes, and self-efficacy mediate any effect of post-lapse patch use on abstinence.
Time Frame: 4 months after the quit date
Population: Because the results for the primary outcome were negative, this outcome was not analyzed (i.e., there was no effect to mediate).
Arm/Group | Nicotine Patch, Experimental Use | Nicotine Patch, Labeled Use
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Adverse Drug Effects
Description: To test whether the incidence of adverse drug effects during the post-lapse use of nicotine patch is minimal.
Time Frame: Up to 12 weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Patch, Experimental Use | Nicotine Patch, Labeled Use
Number analyzed (Participants) | 356 | 345
Participants | 37 | 27
Statistical Analysis 1: Comparison: Nicotine Patch, Experimental Use vs Nicotine Patch, Labeled Use; Comparison of number of participants who reported removing the nicotine patch due to a side effect; Test type: Superiority; p = 0.24, Chi-squared

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Nicotine Patch, Experimental Use | Nicotine Patch, Labeled Use
All-Cause Mortality (participants affected / at risk) | 1/356 | 1/345
Serious Adverse Events (participants affected / at risk) | 4/356 | 4/345
Other Adverse Events (participants affected / at risk) | 196/356 | 187/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Patch, Experimental Use (N=356) | Nicotine Patch, Labeled Use (N=345)
Stroke (Vascular disorders) | 0 | 1
Intestinal problems (Gastrointestinal disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Pancreas problems (Endocrine disorders) | 0 | 2
Hospitalization (General disorders) | 2 | 0 — 1 hospitalization and 1 death due to unknown causes
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Patch, Experimental Use (N=356) | Nicotine Patch, Labeled Use (N=345)
Insomnia (Psychiatric disorders) | 79 | 78
Skin irritation (Skin and subcutaneous tissue disorders) | 122 | 120 — Redness or irritation at the patch site
Dizziness (Nervous system disorders) | 33 | 31
Headache (Nervous system disorders) | 44 | 37
Nausea (Gastrointestinal disorders) | 35 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No